CLINICAL TRIAL: NCT04744103
Title: Trichloroacetic Acid as a Topical Treatment for Actinic Cheilitis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: This study has been on hold due to the COVID-19 pandemic. Recruitment never began and the team didn't renew the study
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1026120
Record Dates: First submitted 2021-01-31; First posted 2021-02-08 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Actinic Cheilitis
MeSH Terms: conditions — Actinic cheilitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- TCA peal (Experimental): Patients will have their actinic cheilitis treated with a TCA peal.
  Interventions: Drug: TCA

INTERVENTIONS:
Drug: TCA — Patients will receive a TCA peel as a treatment for their actinic cheilitis.

SUMMARY:
Actinic cheilitis is a condition of the lower lip characterized by grayish-white areas of discoloration and blunting of the demarcation between the cutaneous lip and the mucosa.

While many studies have compared treatment options for actinic cheilitis, there is still significant debate over how to best manage this condition. The chosen treatment regimen must result in complete remission while also preventing recurrence and malignant transformation. Current treatment options are vast, including both non-surgical and surgical options. Common topical therapies include 5-fluorouracil, imiquimod, ingenol mebutate and diclofenac. More recently, photodynamic therapy has been brought forward as a potential treatment modality. From a surgical perspective, a vermilionectomy is typically the procedure of choice.

TCA is a popular topical treatment for treat fine rhytides, hyperpigmentation, photodamage, and premalignant changes, such as actinic keratoses. Despite this, TCA is not commonly used for actinic changes on the lips. Here, the investigators propose an expansion of the application of TCA to be used in the treatment of actinic cheilitis.

DETAILED DESCRIPTION:
The proposed study will be a prospective cohort study of all patients with actinic cheilitis presenting to the study institution, the Queen Elizabeth II Health Science Center in Halifax, from March 1st 2021- March 1st 2023.

Patients will be consented to participate at the time of their initial consultation. They will fill out the demographics form, a preliminary survey and have the required photographs taken on that same day. A biopsy will be performed prior to treatment to establish the histological grade of their actinic cheilitis based on the degree of dysplasia. After the treatment is received, they will follow-up in 1 month for reassessment. At this point, a second treatment will be offered if clinical remission has not been achieved. Patients will continue TCA treatments at 1-month intervals until clinical remission is reached. Once remission is achieved, they will fill out the post-treatment questionnaire and have their second set of photos taken.

Final follow-up will occur 6 months post remission. At this point patients will be assessed for clinical recurrence. A third set of photos will be completed during this appointment.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will include all patients with actinic cheilitis that do not meet exclusion criteria.

Exclusion Criteria:

* Exclusion criteria will include patients younger than 18 years of age and patients with a biopsy proven malignancy of the lip.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Remission rate | 3 months
  Determine the remission rate of actinic cheilitis following topical TCA treatment.
Treatment Number | 3 months
  Establish the average number of treatments required to achieve remission.
Recurrence Rate | 6 months
  Determine the recurrence rate of actinic cheilitis following topical TCA treatment
Adverse Events | 3 months
  Identify the common adverse events, if any, associated with topical TCA lip peels and determine their incidence.

SECONDARY OUTCOMES:
patient satisfaction | 6 months
  Identify patient satisfaction before and after TCA treatment using the Skindex 16 survey developed by the University of California. This survey looks at how bothered patients are by a skin condition, with a higher score representing a more severe condition. The survey will be completed before and after treatment and the improvement in the score will be analyzed. There are 16 questions, each with a max score of 6, making the total survey score out of 96 and a minimum score of 0. A higher score indicates a poor quality of life attributed to the described skin condition.
Healing Time | 6 months
  Determine the average healing time following TCA lip treatments- self reported

CONTACTS AND LOCATIONS:
Locations (1):
- QEII, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
Participant data will not be used outside the confines of this study.

REFERENCES:
- [Derived] Kuta V, Taylor SM. Trichloroacetic Acid as a Topical Treatment for Actinic Cheilitis. OTO Open. 2025 May 23;9(2):e70132. doi: 10.1002/oto2.70132. eCollection 2025 Apr-Jun. PMID 40416781